CLINICAL TRIAL: NCT01630382
Title: Cerebrospinal Fluid Congestion in Spinal Stenosis Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: H-1203-088-402
Record Dates: First submitted 2012-06-26; First posted 2012-06-28 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2012-06

CONDITIONS: Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators hypothesized spinal stenosis symptom was provocation due to cerebrospinal fluid congestion.

ELIGIBILITY:
Inclusion Criteria:

* neurogenic claudication more than 3months
* relief neurogenic claudication by lumbar flexion
* spinal stenosis symptom by physical exam.
* who can walk more than 30 min.

Exclusion Criteria:

* vascular claudication by physical exam.( ABI <0.9)
* structural change in vertebral ( tumor, congenital deformity)
* operation history at spinal bone
* metallic foreign body
* peripheral polyneuropathy

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: study group : spinal stenosis patient control group : matched sex, age
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2012-06; Primary Completion 2013-05 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
CSF pressure at spinal canal | on time of recruitment
  We can calculate CSF pressure at spinal canal by using phase contraast magnetic resonance image technique.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea